CLINICAL TRIAL: NCT03334097
Title: Educational Intervention in the Fear-Avoidance Delivery: a Prospective Study.
Brief Title: Educational Intervention in the Fear-Avoidance Delivery
Acronym: FADel_edu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Principal Researcher CTS631, University of Malaga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMA - 2017_FAD
Record Dates: First submitted 2017-07-12; First posted 2017-11-07 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2017-05

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; fear; Parturition; Prenatal Education
MeSH Terms: interventions — Prenatal Education

STUDY DESIGN:
Intervention Model Description: A single groupof pregant women will complete the spanish version of Delivery Expectancy/Experience Questionnaire, Version A (WDEQ-A, spanish version) before and after an educational information.
Masking Description: There will be no masking as the purpose of the study is to analyse responsiveness of a questionnaire after educational intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): There will only one experimental arm in order to study test-retest validity after having validate the questionnaire. The beginning of the maternal education takes place between 26 and 30 weeks of gestation and ends between 32 and 36 weeks of gestation. Hence, to study responsiveness, questionnaires will be filed at the beginning of the maternal education and after the two educational sessions related to childbirth.
  Interventions: Other: Prenatal education

INTERVENTIONS:
Other: Prenatal education — Education intervention will consist of a total of six sessions one week apart, with two hours of duration each one. The sessions that are exclusively oriented towards preparation for childbirth are session 1 and session 2. The content of each session is:
  1. St. Birth: Start of childbirth, Symptoms and Signs, Delivery schedules, Phases of childbirth, Normal childbirth, Other circumstances (Obstetrical pathology / previous pathology, Induction of labor, Instrumental birth, Caesarean section).
  2. nd:methods for relieving birth pain: Alternative Methods of Pain Relief, Pharmacological analgesia, Regional analgesia. Local and regional anesthesia, General anesthesia, breathing training and accompaniment during childbirth-
  3. rd: Puerperium.
  4. rd :Breastfeeding
  5. rd : Newborn care
  6. rd :Positive parenting.

SUMMARY:
The aim of this research is to study the responsiveness of the Spanish Version of Wijma Delivery Expectancy/Experience Questionnaire, Version A (WDEQ-A) in pregnant women after an educational intervention.

DETAILED DESCRIPTION:
The Wijma Delivery Expectancy/Experience Questionnaire is a self-report instrument designed to measure the fear of childbirth in terms of the woman's cognitive appraisal of childbirth, which is now the most commonly used measure of fear of childbirth. The version A, measures the fear before a delivery (WDEQ-A). It consists of 33 items on a 6-point Likert scale (0 = do not agree; 5 = totally agree). The total score ranges from 0 to 165; the higher the score, the greater the fear the pregnant women experience. A higher score (over 85) indicates a more intense fear of childbirth, and a score of over 100 is considered as a phobia; thus, the scale can measure individual degrees of fear among women before and after their deliveries In Spain, there is no specific instrument to test the effectiveness of different practices that are commonly used to reduce the fear of childbirth as the maternal education. Hence, after cross-cultural adaptation into Spanish of the questionnaire (WDEQ-A-Sp), the responsiveness after and educational intervention will be analysed.

Descriptive analyses will be applied to calculate means and standard deviations of the demographic variables. Distribution and normality will be determined by the one-sample Kolmogorov-Smirnov tests (significance >0.05). Responsiveness will calculated following COSMIN requirements.

ELIGIBILITY:
Inclusion Criteria:

* Spanish women living in Málaga, > 18 years old, 26-30 weeks pregnant, to fill all the items of the questionnaires, to perform sessions the Maternal Education Protocol in Malaga

Exclusion Criteria:

* No performin inclusion criteria. No voluntary participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Responsiveness of WDEQ-A-Sp after an educational intervention | inmediate effect
  Responsiveness of Spanish Version of Wijma Delivery Expectancy/Experience Questionnaire, Version A (WDEQ-A-Sp) after an educational intervention in pregnant women

SECONDARY OUTCOMES:
Age | baseline, inmediate effect and 2,4 and 12 weeks. Long time effect 6 months
  Age expressed in years
Weight | baseline, inmediate effect and 2,4 and 12 weeks. Long time effect 6 months
  Weight expressed in kilograms (Kg)
Height | baseline
  Stature expressed in meters (m)
Body Mass Index | aseline, inmediate effect and 2,4 and 12 weeks. Long time effect 6 months
  Body Mass Index (BMI) expressed in kilograms per square meter (Kg/m2)
Educational level | baseline
  Education qualification: Junior high school, High School or Degree/Master degree
Weeks of gestation | baseline
  Weeks of gestation at the start of the study expressed in numbers
civil status | baseline
  Marital status: married/ stable couple; Inestable couple; single
Obstetric history | baseline
  Obstetric information if there have been previous birth(s): No pregnancy, Natural birth, natural with with epidural, instrumental delivery, cesarean operation or emergency cesarean operation
evolution of pregnancy | baseline, inmediate effect and 2,4 and 12 weeks.
  Current pregnancy risk: low risk, medium risk or high risk
Previous experience of pregnancy | baseline, inmediate effect and 2,4 and 12 weeks.
  No experience, miscarriage or death

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Cuesta-Vargas, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wijma K, Wijma B, Zar M. Psychometric aspects of the W-DEQ; a new questionnaire for the measurement of fear of childbirth. J Psychosom Obstet Gynaecol. 1998 Jun;19(2):84-97. doi: 10.3109/01674829809048501. PMID 9638601
- [Background] Korukcu O, Kukulu K, Firat MZ. The reliability and validity of the Turkish version of the Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) with pregnant women. J Psychiatr Ment Health Nurs. 2012 Apr;19(3):193-202. doi: 10.1111/j.1365-2850.2011.01694.x. Epub 2012 Jan 20. PMID 22260727
- [Background] Pallant JF, Haines HM, Green P, Toohill J, Gamble J, Creedy DK, Fenwick J. Assessment of the dimensionality of the Wijma delivery expectancy/experience questionnaire using factor analysis and Rasch analysis. BMC Pregnancy Childbirth. 2016 Nov 21;16(1):361. doi: 10.1186/s12884-016-1157-8. PMID 27871320
- [Background] Mokkink LB, Terwee CB, Patrick DL, Alonso J, Stratford PW, Knol DL, Bouter LM, de Vet HC. The COSMIN study reached international consensus on taxonomy, terminology, and definitions of measurement properties for health-related patient-reported outcomes. J Clin Epidemiol. 2010 Jul;63(7):737-45. doi: 10.1016/j.jclinepi.2010.02.006. PMID 20494804